CLINICAL TRIAL: NCT05981586
Title: Comparative Effects of Plyometric and Isotonic Strengthening Exercises on Speed, Agility and Balance of Lower Extremity Among Field Tennis Players
Brief Title: Comparative Effects of Plyometric and Isotonic Strengthening Exercises of Lower Extremity Among Field Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: REC/RCR&AHS/23/0415 Muneeb
Record Dates: First submitted 2023-04-18; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Lower Extremity Problem
Keywords: Agility, Balance, Isotonic, Plyometric, Tennis players

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPEED (Experimental): Speed tests are typically used solely to measure an athlete's linear speed capabilities. Track sprinters have been shown to accelerate continuously through at least 50m during a 100m sprint event.
  Interventions: Other: Plyometric strengthening exercises; Other: Isotonic strengthening exercises
- BALANCE (Experimental): The person performing the test must maintain their balance on one leg, while using the other leg to reach as far as possible in 8 different directions. The person (standing on his/her left leg for example) must reach in 8 different positions, once in each of the following directions: anterior, antero medial, medial, posteromedial, posterior, posterolateral, lateral and anterolateral.
  The reliability of the SEBT as being moderate to good
  Interventions: Other: Plyometric strengthening exercises; Other: Isotonic strengthening exercises
- AGILITY (Experimental): The T-Test is one of the most important agility Test, used in a lot of different sports all around the world. The test is a combination of different sport specific pattern as forward, lateral, and backward movements
  Interventions: Other: Plyometric strengthening exercises; Other: Isotonic strengthening exercises

INTERVENTIONS:
Other: Plyometric strengthening exercises — Comparative effects 1
Other: Isotonic strengthening exercises — Comparative effects 2

SUMMARY:
The Study design will be randomized clinical trial.This study will be conducted in Pakistan Sports Board, Lahore. The study will be completed within duration of eight to ten months after the approval of synopsis. Sample size will be thirty tennis players.Non-probability Convenient sampling will be used to recruit the individuals for the study and then the randomization will be done by lottery method to divide the individuals into two strengthening exercise group. One group is given Plyometric strengthening exercise plan for 5 weeks along with Tennis specific training and on the other hand isotonic strengthening exercise plan for 5 weeks with Tennis specific training and after that their pre and post values will be measured on SPSS version 25. The objective of this study is to Determine Comparative Effects of Plyometric and Isotonic Strengthening Exercises on Speed, Agility and balance of lower extremity among field Tennis Players

DETAILED DESCRIPTION:
The Study design will be randomized clinical trial. This study will be conducted in Pakistan Sports Board, Lahore. The study will be completed within duration of 10 months after the approval of synopsis. Sample size will be thirty tennis players. Non-probability Convenient sampling will be used to recruit the individuals for the study and then the randomization will be done by lottery method to divide the individuals into two strengthening exercise group. One group is given Plyometric strengthening exercise plan for 5 weeks along with Tennis specific training and on the other hand isotonic strengthening exercise plan for 5 weeks with Tennis specific training and after that their pre and post values will be measured on SPSS version 25. The objective of this study is to Determine Comparative Effects of Plyometric and Isotonic Strengthening Exercises on Speed, Agility and balance of lower extremity among field Tennis Players To move around the court swiftly and effectively, tennis players need to be very agile and balanced. Plyometric exercises can help tennis players develop explosive power and speed. Rapid muscle contractions during plyometric exercises can help with acceleration, power, and reaction time. Tennis players can benefit from plyometric exercises like jump squats, box jumps, and medicine ball throws. Tennis players can enhance their range of motion and lower their risk of injury by engaging in flexibility exercises. Yoga, Pilates, and stretching routines can increase flexibility and assist athletes keep their balance and posture while playing For tennis players, isotonic exercises are a crucial part of a successful fitness regimen. Exercises that are isotonic can increase muscle strength and endurance, which is important for generating power in shots and keeping proper posture on the court. Bicep curls, triceps extensions, and lunges are a few isotonic exercises for tennis players. Tennis players must also engage in plyometric exercises because they can enhance their explosive power and quickness. Rapid muscle contractions during plyometric exercises can help with acceleration, power, and reaction time. Tennis players can benefit from plyometric exercises like jump squats, box jumps, and medicine ball throws Tennis players can potentially lower their risk of injury by engaging in isotonic activities. Isotonic workouts can lower the incidence of common tennis injuries like shoulder, knee, and ankle sprains by enhancing muscle strength and joint stability.

Tennis players might benefit from plyometric training to increase their balance and agility. Plyometric exercises feature quick changes in direction and rapid movements, which can help players move more quickly and effectively around the court.

Tennis players that incorporate isotonic and plyometric workouts into their training regimen can enhance their overall performance. Tennis players may hit the ball harder, move around the court more quickly, and enhance their overall performance by developing their strength, power, speed, and agility

ELIGIBILITY:
Inclusion Criteria:

* Racquet Sports Athletes (Tennis,Badminton,Squash,Table Tennis)
* Both Right and Left handers are included

Exclusion Criteria:

* Lower Extremity Injuries (Fractures,Achilles Tendinitis,Muscle Strain etc)
* Lower Extremity Deformities
* Other Systemic Disorders
* Cricket Players
* Sprinters

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
T-TEST | 8 WEEKS
  The Agility T-test is commonly used to assess the ability of team sport athletes to change direction, including acceleration, deceleration, and lateral movement during testing protocols
STAR EXCURSION TEST | 8 WEEKS
  The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals.
20M SPRINT TEST | 8 WEEKS
  Speed tests are typically used solely to measure an athlete's linear speed capabilities. Track sprinters have been shown to accelerate continuously through at least 50m during a 100m sprint event.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No